CLINICAL TRIAL: NCT01442259
Title: An Open-label, Parallel-group Study to Determine the Pharmacokinetics of a Single Dose of AFQ056 in Subjects With Mild, Moderate or Severe Renal Impairment Compared to Age, Sex, and Body Weight-matched Healthy Subjects
Brief Title: An Open-label, Parallel-group Study to Determine the Pharmacokinetics of a Single Dose of AFQ056 in Subjects With Renal Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CAFQ056A2124; 2010-022738-94 (EudraCT Number)
Record Dates: First submitted 2011-09-09; First posted 2011-09-28 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2017-02

CONDITIONS: Mild Moderate; or Severe Renal Impairment
Keywords: Renal impairment,; pharmacokinetics,; safety
MeSH Terms: conditions — Renal Insufficiency | interventions — mavoglurant

ARMS (1):
- All study subjects (Experimental)
  Interventions: Drug: AFQ056

INTERVENTIONS:
Drug: AFQ056

SUMMARY:
The aim of this study was to characterize the pharmacokinetics and safety of AFQ056 in subjects with a different degree of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be of non-child bearing potential as defined as postmenopausal females with no regular menstrual bleeding for at least 1 year prior to inclusion
* Body weight: ≥50kg; BMI: 18-34 kg/m2
* Ability to communicate well with the investigator and comply with the requirements of the study.

For subjects with renal impairment only

* No current clinically significant disease (other than renal impairment), except for stable underlying disease that caused renal impairment, as determined by clinical history and physical examination.
* MDRD-calculated eGFR of <90 mL/min/1.73 m2 based on serum creatinine
* Vital signs (after 3 minutes resting measured in the supine position) should be within normal ranges as deemed by the Investigator.

For healthy subjects only

* No current clinically significant disease as determined by clinical history and physical examination.
* MDRD-calculated eGFR of ≥90 mL/min/1.73 m2 based on serum creatinine.
* Vital signs (after 3 minutes resting measured in the supine position) should be within normal ranges as deemed by the Investigator.

Exclusion Criteria:

* Pregnant or nursing (lactating) females
* Use of any prescription or over-the-counter (OTC) drugs, herbal (e.g. St. John's wort) ordietary supplements (e.g. broccoli, vitamins) within three weeks or five half lives(whichever is longer) prior to dosing with AFQ056 until study completion. This does not include drugs that are used as (symptomatic) treatment of renal impairment (e.g. antihypertensive and antidiabetic drugs) provided such drugs are:

  * used at the same dose within three weeks or five half lives (whichever is longer) prior to dosing with AFQ056 until study completion.
  * not known as inhibitors or inducers of CYP1A1, 1A2, 2C8, 2C9, 2C19, 3A4, 3A5 gp).
* Participation in any clinical investigation or use of any investigational drug within 30 days or five (5) half-lives of a given investigational drug (whichever period is longer); or longer if required by local regulations prior to screening until study completion
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* History of renal transplantation
* History or presence of prolonged QTc interval (males: >450ms; females: > 470 ms), 2nd or 3rd degree AV-block or any other clinically significant ECG abnormalities as determined by medical history and 12-lead ECG recordings at screening and baseline 1.
* History or presence of any clinically significant disease of any major system organ class, within the past 2 years prior to screening, except for renal impairment and underlying diseases causing renal impairment for the subject belonging to the renal impairment groups.
* Subjects undergoing any method of dialysis (hemodialysis or peritoneal dialysis)
* History of or ongoing active substance abuse (including alcohol) within the past 2 years.
* Smokers (use of tobacco products in the previous 3 months). Urine cotinine levels will be measured during Screening and at Baseline for all subjects. Smokers will be defined as any subject who reports tobacco use and/or who has a urine cotinine ≥ 500 ng/mL at screening

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Measure: Area under the plasma concentration-time curve from time zero to infinity (AUCinf) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: Area under the curve from time zero to the last measurable concentration sampling time (Tlast) [mass x time x volume-1] (AUClast) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: Maximum observed plasma concentration (Cmax) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: Terminal elimination half-life (T1/2) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: The apparent systemic (or total body) clearance from plasma following extravascular administration [volume / time] (CL/F) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: The apparent volume of distribution during the terminal elimination phase following oral administration [volume] (Vz/F) | 0, 0.5, 1, 2, 3, 4, 6, 12, 24, 36, 48, 72 hours post dose
Measure: Amount of drug excreted into the urine from time zero to time't' where t is a defined time point after administration [mass units or % of dose] (Ae0-t) | 4 days
Measure: The renal clearance from plasma [volume / time] (CLr) | 4 days

SECONDARY OUTCOMES:
Physical examination | Screening, Day -1, Day 8 +/- 2 days
Measure: Vital signs and body measurements | Screening, Day -1, Day 1, Day 8 +/- 2 days
Measure: ECG | Screening, Day -1, Day 1, Day 8 +/- 2 days
Measure: pulse oximetry | Screening, Day -1, Day 1, Day 8 +/- 2 days
Measure: hematology | Screening, Day -1, Day 4, Day 8 +/- 2 days
Measure: blood chemistry | Screening, Day -1, Day 2, Day 4, Day 8 +/- 2 days
Measure: urinalysis | Screening, Day -1, Day 4, Day 8 +/- 2 days
Measure: AE (adverse events) monitoring | During the study (up to 10 days)
SAE (serious adverse events) monitoring | During the study (up to 10 days) and up to 30 days after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Kiel, Germany

REFERENCES:
- See also: Results for CAFQ056A2124 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6624